CLINICAL TRIAL: NCT04988698
Title: Factors Predicting the Duration of Effectiveness of Viscosupplementation in Knee Arthosis
Acronym: PRESAGE
Status: Completed | Type: Observational
Sponsor: Hopital Nord Franche-Comte (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-A00773-38
Record Dates: First submitted 2021-07-15; First posted 2021-08-03 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Knee Osteoarthritis
Keywords: viscosupplementation
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: none intervention — none intervention

SUMMARY:
Knee osteoarthritis is a frequent condition whose prevalence is estimated at 7.6% of the French population aged 40 to 75, or approximately 2 million individuals . Viscosupplementation (VS) is a symptomatic treatment of knee osteoarthritis recommended by a large number of learned societies. It consists of the intra-articular injection (IA) of hyaluronic acid (HA), to reduce knee pain by restoring normal joint homeostasis impaired by endogenous HA deficiency.

The IA administration of HA can be performed using 2 protocols: repeated weekly injections (3, sometimes 5 injections) and single injections. To date and there is no argument to favor either protocol. Regardless of the formula used, the safety of HA is excellent (RR of adverse reaction versus saline = 1.01, 95% CI 0.96-1.07, P = 0.6). The indication for viscosupplementation is the symptomatic treatment of mild to moderate knee osteoarthritis after failure and / or intolerance of analgesics or nonsteroidal anti-inflammatory drugs (NSAIDs). In this indication, after HA injection the responder rate is in the order of 70% to 75% at 6 months and approximately 50% at 12 months. However, the predictors of the duration of effectiveness of SV are still unknown. The objective of the study is to research the factors influencing the duration of the effectiveness of SV, under real life conditions.

ELIGIBILITY:
Inclusion Criteria:

* All adult outpatients, of both sexes, regardless of age, with a doctor-accepted diagnosis of knee OA and who have been treated with SV within the past 3 years

Exclusion Criteria:

* Patients who have not been treated with SV in the past 3 years.
* Patients who have been treated with VS for an indication other than osteoarthritis of the knee.
* Patients in whom the assessment could not be performed reliably

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A questionnaire is administered by the investigator during the medical consultation. No act is performed outside of patient care.
Sampling Method: Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
Investigate the factors influencing the duration of the effectiveness of SV, under real-life conditions | At inclusion
  Duration (in weeks) during which the patient was satisfied with the treatment

SECONDARY OUTCOMES:
Research for predictive factors will be carried out on the duration of satisfaction | At inclusion
  Research for predictive factors will be carried out on the duration of satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Nord Franche-Comté, Trévenans, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Perruchet S, Balblanc JC, Rapp C, Bourgoin C, Guillochon C, Lohse A, Conrozier T. The Association between Radiographic Features and the Duration of Effectiveness of a Single Injection of Extended-Release Hyaluronic Acid (HANOX-M-XL) in Patients with Knee Osteoarthritis: Preliminary Results of a Prospective Trial. Cartilage. 2023 Jun;14(2):136-143. doi: 10.1177/19476035221109230. Epub 2022 Dec 17. PMID 36527367